CLINICAL TRIAL: NCT04094948
Title: Phase II Clinical Trial of Clenbuterol in Adult Patients With Pompe Disease Stably Treated With Enzyme Replacement Therapy
Brief Title: Phase II Clinical Trial of Clenbuterol in Adult Patients With Pompe Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: hasn't got the funding
Sponsor: Duke University (Other)
Responsible Party: Principal Investigator, Dwight Koeberl, M.D., Ph.D., Professor of Pediatrics, Duke University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00102462
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Pompe Disease (Late-onset)
Keywords: Pompe disease; LOPD; Late-onset Pompe Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — Clenbuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- clenbuterol (Experimental): The initial dose of clenbuterol will be 40 mcg per oral each morning for one week, followed by 40 mcg twice per day (BID) for the next 5 weeks until Week 6. If the 40 mcg BID per oral is well tolerated, the dose will be increased to 80 mcg each morning/40 mcg each evening for one week, followed by 80 mcg BID for the next 5 weeks until the Week 12 visit. If 80 mcg BID is tolerated at Week 12, the subject will continue on that dose until Week 52.
  Interventions: Drug: Clenbuterol
- placebo (Placebo Comparator): Initially, one capsule each morning for one week, followed by one capsule BID for the next 5 weeks until Week 6. If tolerated, the dose will be increased to two capsules each morning and 1 capsule each evening for one week, followed by two capsules BID for the next 5 weeks until the Week 12 visit. If two capsules BID is tolerated at Week 12, the subject will continue on that dose until Week 52.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Clenbuterol — 20 mcg spiropent tablets will be overencapsulated (two 20 mcg tablets per capsule)
  Other Names: Spiropent
  Arms: clenbuterol
Drug: Placebos — dextrose-filled capsules
  Arms: placebo

SUMMARY:
The goals of this study are to determine safety and efficacy with regard to motor function of oral clenbuterol in combination with ERT in subjects with LOPD

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Pompe disease by blood Acid alpha-glucosidase (GAA) assay and GAA gene sequencing,
2. Age: 18+ years at enrollment,
3. Receiving enzyme replacement therapy (ERT) at a stable dose for >104 weeks,
4. FVC >15% of expected (supine).
5. Subjects are capable of giving written consent.
6. Able to walk at least 100 meters on the 6 minute walk test (6MWT) (with assistive devices permitted).

Exclusion Criteria:

1. Continuous invasive ventilation (via tracheostomy or endotracheal tube)
2. 6MWT distance >90% of expected performance (% expected)
3. FVC >90% of expected (upright).
4. Clinically relevant illness within two weeks of enrollment including fever > 38.2o C, vomiting more than once in 24 hours, seizure, or other symptom deemed contraindicative to new therapy.
5. Chronic heart disease (Myocardial infarction, arrythmia, cardiomyopathy)
6. Tachycardia
7. History of seizure disorder
8. Hyperthyroidism
9. Pheochromocytoma
10. Pregnancy
11. History of diabetes
12. History of hypersensitivity to β2-agonist drugs such as albuterol, levalbuterol (Xopenex), bitolterol (Tornalate), pirbuterol (Maxair), terbutaline, salmeterol (Serevent),
13. Patients on a non-standard schedule for ERT; for example, weekly infusions as opposed to infusions every two weeks.
14. Treatment for asthma in the previous 12 months.
15. Renal insufficiency (elevated serum creatinine).
16. Having started respiratory muscle strength training in the last 6 months prior to study day 1 or having discontinued respiratory muscle strength training in the 6-month period preceding study day 1, or having started respiratory strength training greater than 6 months prior to study day 1 and unwilling to continue for the first year of study participation.
17. Received an investigational drug or participated in another interventional study within 90 days of Study Day 1.
18. Anti-rhGAA IgG with sustained titer >1:25.600 for >6 months at time of enrollment.
19. The use of the following concommitant meds is prohibited during the study:

    * diuretics (water pill);
    * digoxin (digitalis, Lanoxin);
    * beta-blockers such as atenolol (Tenormin), metoprolol (Lopressor), and propranolol (Inderal);
    * tricyclic antidepressants such as amitriptyline (Elavil, Etrafon), doxepin (Sinequan), imipramine (Janimine, Tofranil), and nortriptyline (Pamelor);
    * Monoamine oxidase (MAO) inhibitors such as isocarboxazid (Marplan), phenelzine (Nardil), rasagiline (Azilect), selegiline (Eldepryl, Emsam), or tranylcypromine (Parnate); or
    * other bronchodilators such as albuterol, levalbuterol (Xopenex), bitolterol (Tornalate), pirbuterol (Maxair), terbutaline (Brethine, Bricanyl), salmeterol (Serevent), isoetherine (Bronkometer), metaproterenol (Alupent, Metaprel), or isoproterenol (Isuprel Mistometer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in 6 minute walk test (MWT) distance | Baseline (week 0) through 52 weeks

SECONDARY OUTCOMES:
Changes in pulmonary function tests: forced expiratory volume in 1 second (FEV1) | Baseline (week 0) through 52 weeks
Changes in pulmonary function tests: forced vital capacity (FVC) | Baseline (week 0) through 52 weeks
Changes in pulmonary function tests: maximum expiratory pressure (MEP) | Baseline (week 0) through 52 weeks
Changes in pulmonary function tests: Maximum inspiratory pressure (MIP) | Baseline (week 0) through 52 weeks
Changes in graded functional test: Gait, Stairs, Gower, Chair (GSCS) | Baseline (week 0) through 52 weeks
Changes in graded functional test: Quick Motor Function Test (QMFT) | Baseline (week 0) through 52 weeks
Changes in the concentration of alanine transaminase (ALT) in serum | Baseline (week 0) through 52 weeks
  Avoidance of liver toxicity as defined by a a persistent (sustained >2 weeks) >3x increase in aspartate aminotransferase (AST) or alanine aminotransferase (ALT) from the respective baseline values and/or an increase in direct, indirect or total bilirubin of >3x the upper limit of normal (no liver toxicity has been reported in association with clenbuterol administration and therefore repeat testing should be acceptable)
Changes in the concentration of creatine kinase (CK) in serum | Baseline (week 0) through 52 weeks
  Avoidance of Worsening muscle involvement (i.e. muscle weakness, cramping, or fatigue) accompanied by a persistent (sustained >2 weeks) >3x increase in CK from baseline that is >2x the upper limit of normal (elevated CK is associated with LOPD and minor elevations of CK have been reported in association with clenbuterol administration, therefore repeat testing should be acceptable).
Changes in the concentration of urinary glucose tetramer (Glc4) | Baseline (week 0) through 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dwight Koeberl, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No